CLINICAL TRIAL: NCT04801654
Title: A Monocentric, Prospective Clinical Survey on Long Term Performance of GMK Sphere Total Knee Arthroplasty
Brief Title: GMK Sphere TiNb Total Knee Arthroplasty PMS Study
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P.02.01.427
Record Dates: First submitted 2020-12-16; First posted 2021-03-17 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Ion released group: First 30 patients will be assessed for metalic ion released by blood sample. the patients will be monitored until 10 years follow-up for long term performance of the device
  Interventions: Diagnostic Test: blood sample
- Other group: The remaining 125 patients will be not assessed for metalic ion released; they will be monitored until 10 years follow-up for long term performance of the device

INTERVENTIONS:
Diagnostic Test: blood sample — preoperative and at 6 months and 1 year follow-up after the surgery the patients will take a blood sample
  Groups: Ion released group

SUMMARY:
Total knee arthroplasty (TKA) is one of the success stories of modern surgery, providing high patient satisfaction outcomes. Total knee prostheses are generally composed by a femoral component articulating on a polyethylene insert and a tibial tray.

Recently there has been particular attention on the component material; traditionally femoral components are made of cobalt alloys while tibial baseplates are made, in the great majority of cases, of metallic materials, but also polyethylene versions are available. There has been a degree of acceptance in some countries that metal related pathology may exist as demonstrated by the Australian Arthroplasty register where metal hypersensitivity was reported as the fifth most common cause for revision hip arthroplasty 2012 report, making up for 5.9% of all revisions. The wording was subsequently changed from "metal sensitivity" to "metal related pathology" in the 2014 report with 0.5% of all revision total hip arthroplasties (THA) associated with this term. The same change in terminology was used for TKA with metal sensitivity as a cause for revision in 1.3% of revisions in 2012 and in 2014, 1.8% of revision TKAs attributed to "metal related pathology" . The overall revision rate was 3.45% after 10 years in 396.472 TKAs, suggesting a revision rate of 0.06-0.32% secondary to metal or cement allergies. Up to today there is no question that metallic implants may generate wear debris that cause local reactions. This local reaction is not dose related nor predictable and therefore not purely due to the toxic effect of the debris but possibly due to an immunological host process. Hypersensitivity to metal undoubtedly exists but it cannot be stated at the moment to be an allergic reaction. To prevent issues arising due to metal related pathology, alternative solutions to conventional chrome cobalt material have been proposed, for example ceramic component or implant coating. In particular, TiNbN coating has been proposed by most companies thanks to its excellent biological properties. Preclinical studies have showed a high scratch resistance and low coefficient of friction, more resistance to fretting corrosion, reduction of wear, lower ion release rates and low fatigue cycle, as described in the review of Hove. Clinically, cohort of studies of TiN-coated implants showed an overall survival exceeding 90% with a follow-up of 15 to 77 months and good clinical outcomes. No reports of adverse effects related to TiN coating of CoCrMo knee implants have been showed. There are few studies that compared TiN-coated implants with the same uncoated version. Thienpont, comparing TiN-coated and uncoated CoCrMo implants, showed similar clinical and radiological outcomes at short-term follow up in both patients groups .

Overall we can conclude that in literature no adverse events have been reported concerning the TiNbN coating and in particular it has been showed that the coating doesn't not affect the performance of the device if compared with the same uncoated version.

The aim of this study is to evaluate the long term clinical and radiological performance of GMK Sphere total knee component, coated version.

ELIGIBILITY:
Inclusion Criteria:

* Those older than 18 years old at the surgery time
* those suitable to undergo to a primary total knee arthroplasty for whom the GMK Sphere TiNb coated device will be implanted (according to the label indication/contraindications)
* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to patient's surgery

Exclusion Criteria:

* Those patients with metal implants containing Co, Cr and / or Ni
* Those patients who have had environmental or occupational exposure to toxic metals such as Co, Cr and / or Ni (solvents, industrial paints, welders)
* Those whose mental conditions may compromise their ability to provide informed consent to study participation, ability to complete questionnaires or complete 10-year follow-ups
* Those unable to give their consent to participate in the study or who do not want to participate
* Any condition not mentioned in inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample size calculation has been performed according to one proportion test comparing expected survival at 10 year of 96.3%[5] with the bench mark value defined by ODEP Panel for a total knee arthroplasty at 10 yrs of 90%. With a significance level of 5% and a power of 80%, 141 patients are necessary to show a non-inferiority test. Considering a lost to follow-up rate of 10%, 155 patients will be recruited.
  B. Bordini, C. Ancarani, and D. A. Fitch, "Long-term survivorship of a medial-pivot total knee system compared with other cemented designs in an arthroplasty registry," Journal of orthopaedic surgery and research, vol. 11, no. 1, p. 44, 2016
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2033-02-05 (Estimated); Study Completion 2033-12-05 (Estimated)

PRIMARY OUTCOMES:
Long term performance | 10 years
  Device survival will be assessed by Kaplan Maier curve

SECONDARY OUTCOMES:
Clinical performance | 6 months, 1, 5 and 10 years after surgery
  Clinical performance will be assessed through the NEW KSS score collected during preoperative and follow-up visits. The score is divided in subscale: objective (0-75), Symptoms (0-25), Satisfaction (0-40), Expectation (0-15), Functional Activities (0-30), high scores indicating good outcomes.
Radiological performance | (1, 5 and 10 years after surgery
  standard x-ray exam performed preoperatively and postoperatively before discharge from hospital and during follow-up visits
Retropatellar pain | 6 months and 1, 5 and 10 years after surgery
  Kujala score collected during preoperative visit and follow-up visit. Each scale ranges from 0 to 100 with high scores indicating good outcomes.
Ion release rate | preoperative, 6 months and 1 year visits
  blood level of ions Co, Cr and Ni in a subgroup of 30 patients
Activity level after surgery | 6 months and 1year after surgery
  UCLA Activity score collected during preoperative visit and follow-up visit. 1-10 scale with 1 less active, to 10 more active.
Rate of complications | up to 10 years after surgery
  collection of all adverse events occurred

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi di Milano Sede di via Monreale18 (Istituto Clinico San Siro), Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No